CLINICAL TRIAL: NCT02708407
Title: PD-HF: A Multi-centre Randomised Controlled Trial of Intermittent Peritoneal Dialysis With Icodextrin-based Solutions on Patients With Severe Heart Failure and Stage 3-4 Chronic Kidney Disease
Brief Title: PD-HF: A Trial of Peritoneal Dialysis in Patients With Severe Heart Failure and Chronic Kidney Disease
Acronym: PD-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit adequate number of participants
Sponsor: University of Nottingham (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS project ID: 158992; ref: PG/13/27/29864 (Other Grant/Funding Number: BHF grant)
Record Dates: First submitted 2016-01-18; First posted 2016-03-15 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure; Chronic Kidney Disease
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic | interventions — Peritoneal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peritoneal Dialysis Group (Experimental): These participants will continue to receive standard HF care and Peritoneal Dialysis with a single daily exchange of icodextrin.
  Interventions: Procedure: Peritoneal Dialysis
- Control Group (No Intervention): These participants will continue to receive standard HF care.

INTERVENTIONS:
Procedure: Peritoneal Dialysis — One week after insertion of a PD catheter the intervention group will received a single nightly exchange, using dialysis fluid containing icodextrin; a variable proportion of participants may require a second exchange as directed by the consultant nephrologist as part of routine care. The second exchange would use dialysis fluid containing glucose, not icodextrin. Support and training will be given to each participant by the PD specialist team.
  Arms: Peritoneal Dialysis Group

SUMMARY:
This trial is to establish whether ultrafiltration by peritoneal dialysis is a clinically effective treatment for patients with severe heart failure and moderate chronic kidney disease, thus improving quality of life and symptoms.

DETAILED DESCRIPTION:
The trial is a multi-centre, prospective, randomised, unblended, controlled trial of intermittent PD with a single daily exchange of icodextrin plus best standard care versus best standard care for the treatment of severe HF and moderate CKD. A second exchange with glucose based solution may be given, should it be required in the investigator's/clinician's opinion. Investigators will randomise 130 participants for 32 weeks with randomisation stratified by participating centre. Participants will be recruited from specialist-led outpatient HF services in 6 NHS trusts and be managed by both cardiologists and nephrologists.

PD catheter insertion will occur according to the participating centre's institutional protocol. Treatment begins 1 week after catheter insertion and consists of a single nightly exchange.

ELIGIBILITY:
Inclusion Criteria:

* Severe heart failure (NYHA grade III or IV)
* Chronic kidney disease stage 3-4
* Fluid overload resistant to diuretics OR hospital admission for HF in last 6 months
* Left ventricular ejection fraction ≤40% in last 2 years (moderate/severe)
* Using optimal HF medication for ≥ 4 weeks including ACE-inhibitor (angiotensin-converting-enzyme inhibitor) OR angiotensin receptor blocker AND aldosterone antagonist AND beta-blocker unless intolerant and without dose change for ≥ 4 weeks
* Appropriately screened for revascularization and/or cardiac resynchronization therapy if clinically indicated.

Exclusion Criteria:

* Does not wish to participate
* Mental incapacity to consent
* CKD stage 5
* Normal renal excretory function
* Haemodynamically significant valvular disease amenable to surgery
* Cardiac or renal transplantation
* Considered by the investigator to unsuitable for PD due to previous abdominal surgeries, peritonitis, social circumstances or other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The primary end-point is a change of 25 metres walked | Baseline to week 28
  6 Minute Walk Test

SECONDARY OUTCOMES:
Change in KCCQ score | Baseline to week 28
  Kansas City Cardiomyopathy Questionnaire
Change in SF36 score | Baseline to week 28
  Short Form 36 questionnaire
Change in Derby Evaluation of Illness online visual analogue scale | Baseline to week 28
  Derby Evaluation of Illness online visual analogue scale
Heart Failure related hospitalisations | Baseline to week 28
  Recording the number of hospitalisations relating to Heart Failure
All cause hospitalisations | Baseline to week 28
  Recording the number of hospitalisations for all causes
Heart failure related mortality | Baseline to week 28
  Recording the number of heart failure deaths
All cause mortality | Baseline to week 28
  Recording the number of all cause deaths

OTHER OUTCOMES:
Episodes of PD associated peritoneal infection | Baseline to week 28
  Recording the numbers of PD associated peritoneal infections
Adverse events spontaneously reported during the study | Baseline to week 28
  Recording and reporting adverse events
Is the Derby Evaluation of Illness online visual analogue scale more sensitive than pen and ink questionnaires | Baseline to week 28
  Comparison between the scores from pen and ink questionnaires and the online visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Taal, Principal Investigator — University of Nottingham
Locations (1):
- Derby Teaching Hospitals NHS Foundation Trust, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided